CLINICAL TRIAL: NCT01599247
Title: Natural History of Hopelessness, Suicidality, and Optimism in Psychiatric Inpatients Following Discharge
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Medical Director, Blake 11, Massachusetts General Hospital
Other Study IDs: 2010P002851
Record Dates: First submitted 2012-05-02; First posted 2012-05-15 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Suicide, Attempted; Suicidal Ideation
Keywords: Suicide; Optimism; Hopelessness
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suicidal ideation/behavior

SUMMARY:
Specific aim #1: To assess the study team's ability to recruit subjects in this cohort and to successfully complete follow-up assessments by phone or mail.

Hypothesis: Over 50% of eligible subjects will enroll in the observational study, and 70% of follow-up assessments will be successfully completed.

Specific aim #2: To determine the natural history of hopelessness, ongoing suicidal thoughts, and optimism in subjects at 2, 4 and 8 weeks after discharge.

Hypothesis: Subjects will continue to have moderate levels of hopelessness, suicidal thoughts, and optimism at follow-up assessments.

DETAILED DESCRIPTION:
Contact information. On the day of enrollment, contact information (address, phone number) will be obtained from the subject. Subjects will also be asked to provide the contact information for a family member or friend who the study team may contact in case of emergency or if unable to get in touch with subject at follow up. Subjects unable to provide contact information for at least one family member will not be enrolled.

Baseline evaluation.

On the date of enrollment, study staff will obtain two types of information:

1. Baseline clinical characteristics. Study staff will obtain specific clinical variables from the patient to gather information about variables that could impact levels of hopelessness/optimism after discharge. These variables include: age, gender, # of prior admissions [zero, 1-5, more than 5], presence of substance use disorder (assessed via inpatient chart review), admission for suicide attempt or suicidal ideation only, and involvement in exercises that can increase feelings of well-being like gratitude, forgiveness, using one's personal strengths, and acts of kindness.
2. Baseline outcome measures: Study staff will also administer six instruments:

   * Beck Hopelessness Scale (BHS):14 This is a 21-item scale used to assess feelings of hopelessness.
   * Concise Health Risk Tracking Scale (CHRT):15 This is a 12 item scale used to assess the presence and intensity of suicidal thoughts.
   * Life Orientation Test-Revised (LOT-R):16 This is a 10-item scale that measures optimism (and pessimism).
   * Positive Affect Negative Affect Schedule (PANAS):17 This is a well-validated 20-item self-report measure of more general positive and negative affect.
   * Sheehan Disability Scale:18 This is a 5 item scale used to assess the degree to which the subject's condition or disease (psychological, social, physical) has impacted his or her functioning in daily life.
   * Quick Inventory of Depressive Symptomatology, Self Report (QIDS-SR):19 This is a 16-item questionnaire that assesses the subject's depressive symptoms. It will serve as an additional reliable, valid way to gather information on the subject's mood.

This evaluation should take approximately 20-30 minutes.

Follow-up assessments.

Follow-up assessments will occur by phone or mail at 2 weeks, 4 weeks and 8 weeks. Similar to initial assessments, the follow-up assessments will have two components:

1. Assessment of characteristics: Study staff will inquire about subjects' living situation at discharge (homelessness, living alone), employment/academic status, treatment postdischarge (follow-up with therapist, psychiatrist, PCP, groups, AA/NA, partial hospital programs, and other treatment and forms of peer support), and involvement in exercises that can increase feelings of well-being like gratitude, forgiveness, using one's personal strengths, and acts of kindness.
2. Assessment of study outcomes: Staff will readminister the five measures above, and will also inquire about psychiatric readmissions, suicide attempts, and episodes of self-harm (cutting, burning, banging/hitting body parts, ingesting toxic materials/objects, and other intentional non-suicidal self-harm behaviors). This evaluation should take 20-30 minutes.

ELIGIBILITY:
Inclusion criteria:

* Admission to MGH inpatient psychiatric unit, age 18 and older
* Suicidal ideation reported on admission (suicidal thoughts or active suicidal ideation documented in the admission note) OR admission occurring in context of a suicide attempt
* Mood disorder (assessed and determined by patient's clinical treatment team and consulting inpatient chart review)
* Patient able to read and write in English

Exclusion criteria:

* Psychotic symptoms, as assessed using the MINI12 and inpatient chart review
* Cognitive disorder, as assessed using a six-item cognitive screen developed for research
* Participation in other studies that are focused on improving hopelessness/optimism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Inpatient Psychiatric Unit at Massachusetts General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Ability to recruit and retain subjects in this cohort | 2 years
  Number of subjects who enroll in the study, and number of subjects who complete phone or written follow-ups at each time point.

SECONDARY OUTCOMES:
Change in the natural history of hopelessness, suicidal thoughts, and optimism | 2, 4, and 8 weeks
  Changes in scores between baseline and 2/4/8 weeks after discharge. Rates of readmission to hospital, suicidal thoughts, and non-suicidal self-harming behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States